CLINICAL TRIAL: NCT01988987
Title: Evaluating for Type-2 Diabetes in the Very Early Post-Partum Period
Brief Title: Evaluating for Type-2 Diabetes in the Very Early Postpartum Period
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: WUH 12318; 18-01705 (Other: New York Langone Institutional Review Board)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Diabetes, Gestational; Prediabetic State; Glucose Metabolism Disorders; Diabetes Mellitus
Keywords: Gestational diabetes; Postpartum glucose testing; Impaired glucose metabolism; Diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational; Prediabetic State; Glucose Metabolism Disorders; Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inpatient Postpartum GTT: Women with gestational diabetes will undergo a 75 gram, 2 hour, oral glucose tolerance test 2-4 days postpartum prior to hospital discharge, in addition to undergoing the standard of care, outpatient glucose tolerance test performed 6-12 weeks postpartum
  Interventions: Other: Inpatient Postpartum GTT

INTERVENTIONS:
Other: Inpatient Postpartum GTT — Women with gestational diabetes will undergo a 75 gram, 2 hour, oral glucose tolerance test 2-4 days postpartum prior to hospital discharge, in addition to undergoing the standard of care, outpatient glucose tolerance test performed 6-12 weeks postpartum
  Other Names: Glucose tolerance test; Oral glucose tolerance test; OGTT

SUMMARY:
Pregnancy-associated diabetes, known as gestational diabetes mellitus (GDM), is associated with an increased lifetime risk of developing diabetes mellitus (DM) or pre-diabetes. Up to 30% of women with GDM will continue have abnormal blood glucose tests 6 or more weeks after delivery. Early diagnosis and treatment of continued impaired glucose metabolism or DM is essential because serious health problems can result.

Current guidelines recommend a 75-gram, 2-hour glucose tolerance test (GTT) 6 or more weeks after delivery for women diagnosed with GDM in order to identify those with continued DM or impaired glucose metabolism. However, approximately half of these women do not get glucose testing after delivery. The ability to test women while they are still hospitalized after having a baby could greatly increase diagnosis, care and treatment of women with abnormal glucose metabolism.

Our objective is to determine if a 75-gram, 2-hour GTT administered to women with GDM two to four days after delivery can identify those who will have an abnormal GTT at 6-12 weeks after delivery.

DETAILED DESCRIPTION:
This will be a prospective cohort study conducted at Winthrop-University Hospital. Women 18 years old or older who delivered a child or fetus within the previous 4 days at either hospital who also were diagnosed with GDM during the pregnancy will be eligible for participation. Women will be excluded if they have issues that would interfere with administration of a GTT, are unable /unwilling to provide informed consent, or cannot follow up. Anticipated enrollment will be 250 women at each study site.

While still hospitalized two to four days postpartum, subjects will undergo a 75-gram, 2-hour GTT and have blood tested for hemoglobin A1c and glucose levels. They will be reminded to do the recommended GTT 6-12 weeks after delivery. Maternal, neonatal, and obstetric characteristics will be collected, including the any GTT results. The results of the in-hospital GTT will be compared to the result of the GTT taken 6-12 weeks postpartum and tested for correlation.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years old or older
* Delivered a child or fetus within the previous 4 days
* Diagnosed with gestational diabetes during the pregnancy

Exclusion Criteria:

* Unable or unwilling to provide informed consent for the study
* Unable to undergo or complete a 2-hour oral glucose tolerance test 2-4 days postpartum
* Unable or unwilling to have study follow up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women hospitalized for delivery at a teaching hospital.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Result of an early postpartum 75-gram oral glucose tolerance test (GTT) result | 2-4 days postpartum
  The GTT result obtained 2-4 days postpartum will be compared to the GTT result obtained 6-12 weeks postpartum using the McNemar test for paired proportions.

SECONDARY OUTCOMES:
Result of a postpartum 75-gram oral glucose tolerance test (GTT) | 6 weeks-6 months postpartum
  The GTT result obtained 2-4 days postpartum will be compared to the GTT result obtained 6-12 weeks postpartum using the McNemar test for paired proportions.

CONTACTS AND LOCATIONS:
Overall Officials: Jolene Muscat, M.D., Principal Investigator — NYU Winthrop Hospital
Locations (1):
- NYU Winthrop Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided